CLINICAL TRIAL: NCT02871583
Title: The Evaluation of Trunk Muscle Strength, Quality of Life, and Neuropathic Pain Component After Two Different Inguinal Hernia Repair Techniques; A Prospective Controlled Trial
Brief Title: Effect of Inguinal Hernia Repair on Isokinetic Muscle Strength
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Konya Meram State Hospital (Other)
Responsible Party: Principal Investigator, Barış Sevinç, principle investigator, Konya Meram State Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: izokinetic01
Record Dates: First submitted 2016-08-10; First posted 2016-08-18 (Estimated); Last update posted 2016-08-18 (Estimated); Status verified 2016-08

CONDITIONS: Inguinal Hernia
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- lichtenstein (Active Comparator): lichtenstein procedure
  Interventions: Procedure: lichtenstein
- Kugel (Active Comparator): Kugel procedure
  Interventions: Procedure: Kugel
- control (No Intervention): healthy volunteers

INTERVENTIONS:
Procedure: lichtenstein — tension free mesh hernioplasty (lichtenstein) procedure will be applied for inguinal hernia repair
  Arms: lichtenstein
Procedure: Kugel — preperitoneal mesh hernioplasty (Kugel) procedure will be applied for inguinal hernia repair
  Arms: Kugel

SUMMARY:
The aim of the present prospective controlled study is to compare the trunk muscle strength, quality of life and neuropathic pain component after Lichtenstein and Kugel procedures.

DETAILED DESCRIPTION:
In this study patients underwent inguinal hernia repair will be evaluated for the effect of the surgical procedure on abdominal muscle strength.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Male gender (for minimizing the certain effect of gender to muscle strength)
* Patients aged 18-65 years' old
* Having no previous surgery
* Patients within six months to postoperative first year
* Ability to speak, read, and write Turkish

Exclusion Criteria:

* Infections or tumors of the spine
* Systemic bone or joint disorders (e.g., rheumatoid arthritis)
* Unstable cardiovascular and pulmonary diseases
* Polyneuropathies and musculoskeletal system diseases
* Presence of a diagnosed severe psychiatric disorder
* Presence of severe pain
* Regular exercise habit
* Recurrent operation for a hernia
* Presence bilateral inguinal hernia on concurrent femoral hernia
* If the calculated Body mass index is lower than 20kg/cm2 or over than 35kg/cm2

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-12; Primary Completion 2014-02 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
isokinetic muscle strength | 6 - 12 months
  Trunk muscle strength measurement using the Biodex System 3Pro Multi-joint System Isokinetic dynamometer. Peak torque (PT) and PT-based agonist/antagonist ratios will be used to reveal strength imbalances.

SECONDARY OUTCOMES:
quality of life assesment | 6 -12 months
  Quality of life assesment will be performed by Short Form 36 (SF-36) and The PainDETECT questionnaires (PD-Q).

CONTACTS AND LOCATIONS:
Locations (1):
- Konya Training and Research Hospital, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes